CLINICAL TRIAL: NCT07088991
Title: Clinical and Demographic Characteristics of Adult Patients With NEurofibromatosis in RUSsia
Brief Title: Clinical and Demographic Characteristics of Adult p Atients With NEurofibromatosis in RUSsia
Acronym: NEREUS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D134BR00007
Record Dates: First submitted 2025-07-03; First posted 2025-07-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neurofibromatosis
MeSH Terms: conditions — Neurofibromatoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Clinical and Demographic Characteristics of Adult Patients with NEurofibromatosis in RUSsia (NEREUS)

DETAILED DESCRIPTION:
Open-label single-arm, non-interventional, multi-center, cohort study for evaluation of clinical and patient reported outcomes in routine care settings

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of inclusion.
2. Signed and dated written informed consent in accordance with ICH-GCP and local law prior to inclusion in the study.
3. NF1 diagnosed (according to the international consensus criteria for evaluating NF1 [18]), see Appendix A.
4. Confirmed PN by clinical assessment, USI, MRI, biopsy; one method is sufficient (histologic confirmation of PN is not necessary in the presence of radiographic findings).
5. Existing of PN-associated symptoms.
6. Adult patients (≥18 years) with newly diagnosed PN or established PN naïve to MEK-inhibitor therapy verified by medical records/histories (e.g., prior prescriptions, hospitalization data).

Exclusion Criteria:

1. The participation in any clinical study currently (patients participating in other non-interventional studies may be included);
2. Patients with the evidence of a malignant glioma, malignant peripheral nerve sheath tumor, or other cancer, requiring treatment with chemotherapy or radiation therapy.
3. In the opinion of the investigator the patient is not able to return for follow-up visits or obtain required follow-up studies.
4. Individuals who are pregnant or breast feeding or who become pregnant while enrolled on this trial, if they are unable to undergo radiographic evaluations or MRI scans requested for research purposes, or other studies which might negatively impact on the pregnancy.
5. Prior receipt of any MEK-inhibitor for PN therapy within 4 months before screening or initiation of therapy prior to age 18 verified by medical records/histories (e.g., prior prescriptions, hospitalization data).
6. Patients who modify their index pathogenetic therapy regimen during the study (for example, pathogenetic antitumor therapy of PN; switching to a different therapy), as determined by the investigator at any protocol-specified visit during the a study, will be excluded from the primary efficacy analysis population from the point of modification onward and will not continue study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Age ≥ 18 years at the time of inclusion.
  2. Signed and dated written informed consent in accordance with ICH-GCP and local law prior to inclusion in the study.
  3. NF1 diagnosed (according to the international consensus criteria for evaluating NF1 [18]), see Appendix A.
  4. Confirmed PN by clinical assessment, USI, MRI, biopsy; one method is sufficient (histologic confirmation of PN is not necessary in the presence of radiographic findings).
  5. Existing of PN-associated symptoms.
  6. Adult patients (≥18 years) with newly diagnosed PN or established PN naïve to MEK-inhibitor therapy verified by medical records/histories (e.g., prior prescriptions, hospitalization data).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Age (full years) at the inclusion into the study (date of Visit 1) | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Age (full years) at the primary NF1 diagnosis | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Proportion of men and women | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Body mass index (BMI), kg/m2; | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Body surface area (BSA), m2 | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Proportion of patients with each educational status (higher, secondary special, secondary general); | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Proportion of patients from each residential region (federal district of Russia); | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Other than PN specific NF1 symptoms and manifestations | Day 0 (Visit 1)
  skin symptoms and manifestations, tumor manifestations (except malignancies), neurological and cognitive manifestations, cardiovascular manifestations, endocrine manifestations, orthopedic manifestations (distinctive osseous lesions), ophthalmological manifestations, NF1 mutation, presence of NF1 diagnostic criteria in one of parents) (frequency distribution at baseline)
NF1-associated complications | Day 0 (Visit 1)
  malignancy, hypertension, vasculopathy, bone symptoms, chronic neurological conditions, neuropathy, and pain
Non-specific NF1-comorbidities, coded by MedDRA system organ class (SOC) and preferred term (PT) | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Proportion of patients with various specific and non-specific NF1-comorbidities | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Proportion of patients with various PN-associated symptoms | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Proportion of patients with various ECOG score | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Proportion of patients with various PN locations | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
PN volume (established by MRI) | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Duration of PN symptoms persistence before inclusion into the study | Day 0 (Visit 1)
  to be calculated between the date when initially symptoms of PN appeared and the date of Visit 1
Duration of PN diagnosis before inclusion into the study | Day 0 (Visit 1)
  to be calculated between the date of primary diagnosis of PN and the date of Visit 1
Medical history of PN | Day 0 (Visit 1)
  size, symptoms, previous medical interventions, surgeries or treatments
Previous physical, instrumental and laboratory examination results | Day 0 (Visit 1)
  To achieve the primary objectives of the study the following baseline clinical and demographic characteristics of patients will be collected or evaluated. The term 'baseline' means that the data is obtained at the inclusion into the study (Visit 1) during retrospective data collection from patient medical documentation or via interview with a patient on Visit 1, where applicable.
Amount and duration of hospitalizations associated with NF1 according to the investigator's opinion, collected from the medical history since the date of NF1 diagnosis | Day 0 (Visit 1)
  if applicable, to be calculated in patients with at least one such hospitalization
Degree of disability at baseline | Day 0 (Visit 1)
  if applicable, to be calculated in patients with presence of disability at Visit 1
Changing in disability degree during the study | Day 0 (Visit 1)
  if applicable, to be calculated in patients with presence of disability at Visit 1

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint-Peretsburg
  - Research Site, Samara
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/